CLINICAL TRIAL: NCT00006205
Title: Combining Medications Treatment for Alcoholism
Brief Title: Alcohol Dependency Study: Combining Medication Treatment for Alcoholism
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bankole Johnson (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Bankole Johnson, Chair of Psychiatry and Neurobehavioral Sciences, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIAAAJOH1052207A1; R01AA013964 (NIH)
Record Dates: First submitted 2000-09-11; First posted 2000-09-12 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Alcoholism
Keywords: alcoholism; alcohol addiction
MeSH Terms: conditions — Alcoholism | interventions — Ondansetron; Cognitive Behavioral Therapy; Topiramate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ondansetron (Experimental): Ondansetron + cognitive behavioral therapy
  Interventions: Drug: ondansetron + cognitive behavioral therapy
- Topiramate (Experimental): Topiramate + cognitive behavioral therapy
  Interventions: Drug: topiramate + cognitive behavioral therapy
- Placebo (Placebo Comparator): Placebo + cognitive behavioral therapy
  Interventions: Drug: Placebo + cognitive behavioral therapy
- Ondansetron + Topiramate (Experimental): Ondansetron + Topiramate + cognitive behavioral therapy
  Interventions: Drug: ondansetron + topiramate + cognitive behavioral therapy

INTERVENTIONS:
Drug: ondansetron + cognitive behavioral therapy — ondansetron (4 mcg/kg b.i.d)
  Other Names: Zofran
  Arms: Ondansetron
Drug: topiramate + cognitive behavioral therapy — topiramate (up to 300 mg/day)
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo + cognitive behavioral therapy — placebo
  Other Names: sugar pill
  Arms: Placebo
Drug: ondansetron + topiramate + cognitive behavioral therapy — ondansetron (4 mcg/kg b.i.d) + topiramate (up to 300 mg/day)
  Other Names: zofran, topamax
  Arms: Ondansetron + Topiramate

SUMMARY:
The purpose of this study is to learn whether ondansetron and topiramate either alone or in combination is safe and effective in the treatment of alcohol dependence. This 13 week out-patient clinical trial is randomized, double-blind, and placebo-controlled. There are post-study follow up visits 1, 2 and 3 months after the end of the study. Participants will receive ondansetron and topiramate either alone or in combination or a placebo coupled with psychotherapy.

DETAILED DESCRIPTION:
This study is a 13 week clinical trial. During the 13 weeks participants receive placebo, ondansetron and topiramate alone or in combination. During the 13 weeks participants come to an outpatient clinic to receive the study medication, physical checks, and cognitive behavioral therapy. The duration of the weekly visit is 3 hours. There is a 1, 2, and 3 month post-study follow up visit. Screening for this study is initially done over the telephone and takes 15-20 minutes. If there is nothing found to make someone ineligible to participate, they come to the out-patient clinic for a more thorough in-clinic screening.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of alcohol dependence and drinking greater than or equal to 14 alcohol drinks/week for women and greater than or equal to 21 alcohol drinks/week for men in the last 30 days.
* Provide a written, informed consent.
* Good physical health and must weigh within at least 40 kg and no more than 140 kg.
* Literate in English and able to read, understand, follow instructions, and complete questionnaires accurately.
* Willingness to participate in behavioral treatments for alcoholism.
* Provide evidence of stable residence in the last month prior to enrollment in the study and have no plans to move during the next three months.

Exclusion Criteria:

Please contact site for additional information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2005-03; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Self-report measures of alcohol-related problems and consumption, Objective measures of alcohol consumption | Throughout the study
  Drinks per drinking day, Drinks per day, Percent Days Abstinent, BAC, CDT, GGT

SECONDARY OUTCOMES:
Medication compliance, alcohol craving, social functioning, quality of life, alcohol withdrawal, attendance at psychosocial services, pre-morbid risk factors | Throughout the study
  Pill Count, Q-LES-Q, SFQ, AASE, ADBS, OCDS, CIWA-Ar, CGI, TCI, MAC, AOQ, FHAM

CONTACTS AND LOCATIONS:
Overall Officials: Bankole Johnson, DSc, MD, PhD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia Center for Addiction Research and Education, Charlottesville, Virginia
  - University of Virginia Center for Addiction Research and Education, Richmond, Virginia

REFERENCES:
- [Background] Johnson BA. An overview of the development of medications including novel anticonvulsants for the treatment of alcohol dependence. Expert Opin Pharmacother. 2004 Sep;5(9):1943-55. doi: 10.1517/14656566.5.9.1943. PMID 15330732